CLINICAL TRIAL: NCT04469972
Title: Effect of Breathing Exercise on Certain Physiological Parameters, Sleep Quality and Vitality in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aysun Erdal (Other)
Collaborators: Gazi University (Other)
Responsible Party: Sponsor-Investigator, Aysun Erdal, reseach assistant, Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: not have
Record Dates: First submitted 2020-07-02; First posted 2020-07-14 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Breathing; Sleep Disorder
Keywords: Elderly; Breath exercise; Physiological changes
MeSH Terms: conditions — Respiratory Aspiration; Sleep Wake Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation in the intervention group (Experimental): This group of elderly were subjected to a pursed-lip breathing exercise (using a windmill toy), a diaphragmatic breathing exercise and a coughing exercise three times a week (Mondays, Tuesdays and Thursdays) for 12 weeks in groups of 5-6 individuals (2 groups of 6 persons, and 4 groups of 5 persons: 6 groups in total) between 10:00 and 15:30, at the same time of the day for each group in 30-minute sessions. All breathing exercises were taught to the elderly individuals on the first day of implementation and demonstrated again prior to practice by the researcher throughout the implementation phase.
  Interventions: Other: Breathing Exercises
- Implementation in the control group (No Intervention): None of the elderly in the control group were subjected to breathing exercises. They continued their daily lives as normal.

INTERVENTIONS:
Other: Breathing Exercises — Breathing exercise is defined as therapeutic intervention to create a particular form of breathing.The application of the breathing exercise program is as follows; I. Pursed Lip Breathing Exercise (Total 10 minutes) II. Diaphragmatic breathing exercise (10 minutes in total), III. Cough exercise (Total 10 minutes)
  Arms: Implementation in the intervention group

SUMMARY:
Objective: To determine the effect of breathing exercises on certain physiological parameters, sleep quality and vitality in the elderly. Method: In this randomized controlled, experimental study, pre and post tests were applied to 26 elderly participants in the intervention group and to 25 elderly patients in the control group. The intervention group underwent breathing exercises for 30 minutes at the same time of the day, three days a week for three months (pursed-lip breathing exercise, deep breathing exercise, coughing exercise), while no such exercise was carried out by the control group. Pittsburg Sleep Quality Index, the Subjective Vitality Scale, spirometer, sphygmomanometer and pulse oximetry device measurements were used for the collection of data. The data was evaluated with an independent sample t-test, a paired-sample t-test and a two-way repeated measures ANOVA.

DETAILED DESCRIPTION:
Study design The study was conducted in a pre-test- post-test, randomised controlled (parallel) and experimental design.

Study population and sample The sample size was determined based on the variable under study (i.e. lung function) using the GPower 3.1.9.4 program. The pretest and post-test "FVC (L)" variable values obtained by Jun et al.18 were taken into account in the effect size calculations, being 3.26 and 3.46, with standard deviations of 0.33 and 0.61, respectively. The calculations identified a sample size that provides α = 0.05, and the power of the test (1-β) = 0.80 indicated a sample size of 26 subjects in each group. Considering the potential for losses over the course of such studies,12,15 20% of the minimum sample size (11 individuals) was added to the study so as not to reduce the statistical power of the study. It was planned in the study to include 32 elderly participants in the intervention group and 31 in the control group.The study was completed with 26 individuals in the intervention group and 25 individuals in the control group.

Sampling After the study protocol was approved by the Institutional Ethics Committee of Gazi University and the Ministry of Family and Social Policies, a nursing home selected previously according to the number of elderly people in residence was selected for the study and approached. Of the 294 elderly residents of the nursing home, 158 were excluded for not satisfying the inclusion criteria, while 60 were unwilling to take part. Consequently, 63 elderly people were entered into the study and were randomly assigned to the intervention or control groups. While assessing the residents in terms of the inclusion criteria in the study, their health status was obtained from the health unit files of the nursing home, and the Mini Mental test was applied by the researcher.

Randomisation Age and gender are significant factors affecting lung and cardiac function, and so a stratified randomization was performed to ensure the similarity of the intervention and control groups. The study participants were stratified by age (65-74 years, and ≥75 years) and gender (female/male) by the researcher, and were then assigned to the intervention and control groups using a simple randomization application within the computer-based SPSS program, with each stratum group divided equally. In this way, a balanced distribution of the groups was achieved without being affected by age and gender. Neither the study participants nor the breathing exercise trainers were blinded in the study, although the respiratory function tests were evaluated by an independent physiotherapist. The participants were called in alphabetical name order, and the measurements were made by an independent physiotherapist. The statistical analyses and reporting were performed by an independent statistician. The data were sent to the statistician with the groups coded as "Group 1" and "Group 2", without distinguishing between the intervention and control groups.

Implementation steps Pre-test: The pre-test measurements were performed by the researcher and a physiotherapy specialist in the physical therapy unit of the nursing home. The participants in both groups were called up for pretest evaluation in alphabetical name order. To begin with, the PSQI and SVS were applied by the researcher, after which the height and body weight of the participant were measured and recorded, along with their age. All these measurements take around 15 minutes. In this way, the elderly were rested and prevented from imbibing anything that could affect lung and heart function, such as cigarettes, tea or coffee, before measurement. The cardiological findings were then evaluated by the researcher. A manual sphygmomanometer and a pulse oximeter were used to assess cardiac function (blood pressure, heart rate, oxygen saturation). Prior to the oxygen saturation measurement, any blue, black, green, brown or red nail polish was removed, along with any artificial nails. Finally, pulmonary function was assessed, for which dentures were removed. The pulmonary function test procedure had been explained and shown previously by the physiotherapist to the elderly participant, and a spirometer was used for the pulmonary function (FVC, FEV1, FEV1/FVC ratio and percentages) measurement. The results were all delivered to the researcher by the authorized representative of the spirometer manufacturer in pdf format within 15 days. All other data were recorded by the researcher after measurement.

Implementation in the intervention group: A review of literature was made prior to the determination of the breathing exercise protocol to be applied to the elderly participants in the intervention group. In Jun et al., elderly smokers were given breathing exercises three times a week.18 In the study conducted by El Kader, a breathing exercise program was developed for the elderly participants involving activities three times a week for 20 minutes for a period of three months.21 Jansang et al. devised a three-month breathing exercise program for the elderly comprising a diaphragmatic breathing exercise and a pursed lip breathing exercise.12 The breathing exercises in the present study were planned taking into account the methods and recommendations made in the above and similar studies. The intervention group was subjected to a pursed-lip breathing exercise (using a windmill toy), a diaphragmatic breathing exercise and a coughing exercise, three times a week (Mondays, Tuesdays and Thursdays) for 12 weeks in groups of 5-6 (2 groups of 6 persons, and 4 groups of 5 persons: 6 groups in total) between 10:00 and 15:30, at the same time of the day for each group in 30-minute sessions. The exercises were performed in the group activity hall of the physical therapy unit, which was determined as the most suitable area for the participants and for the exercise application, based on a joint decision of the nursing home management and the researcher. No special clothing or equipment was identified for the breathing exercise. The wind rose to be used during the exercise was provided by the researcher. All of the breathing exercises were taught to the participants on the first day of implementation, and were demonstrated again by the researcher prior to exercising throughout the implementation phase. The participants were informed about the possible symptoms that could occur during the breathing exercise, such as dizziness, and they were told to take a short break in such cases, and to wait until the dizziness was over before continuing. If the elderly person could not participate in the exercise session for any reason, the missing exercise time was compensated for the week and day, determined jointly by the elderly individual and the researcher. The breathing exercise program was as follows:

I. Taking the appropriate position for the exercise, as demonstrated by the practitioner (5 minutes) II. Pursed-lip breathing exercise (using a windmill toy) (10 minutes) III. Take a break for 1 minute IV. Diaphragmatic breathing exercise (10 minutes) V. Take a break for 1 minute VI. Coughing exercise (10 minutes)

Implementation in the control group: None of the participants in the control group were subjected to breathing exercises, and continued their daily lives as normal.

Post-test: On the day following the breathing exercises, the PSQI, SVS and physiological parameters were applied following the same steps as in the pre-test implementation, and conducted by the same physiotherapist and researcher in the physical therapy unit. All data were recorded by the researcher in the same manner.

Data assessment The study data were evaluated using the SPSS (Statistical Package for Social Sciences) 16.0 software package. The normal distribution of the quantitative data was assessed with a Kolmogorov-Smirnov test. Numbers, percentages, means, and standard deviation and t-test values were used for the analysis of the dependent groups, and a paired samples t-test, and two-way analysis of variance was used for repeated measures. The level of significance was accepted as p<0.05. The effect size was determined based on Cohen's d value, and a partial eta square (pη2) was used as the effect size when assessing the two-way analysis of variance.

ELIGIBILITY:
Inclusion Criteria:

* Residing individuals at a nursing home in Ankara included the study;

  * aged 65 years and older
  * had a Mini Mental Test score of ≥24,15
  * had no acute or chronic lung diseases,
  * had no physical/mental disabilities or limitations and conditions that might present any obstacle to participate in breathing exercises.

Exclusion criteria. Physical / mental disability or limitation and disease that will prevent them from participating in breathing exercise (previous ear, brain, spinal cord surgery, acute retinal hemorrhage vertebral fracture and diaphragmatic rupture, hiatus or abdominal hernia, acute myocardial infarction, unstable angina pectoris, severe coronary artery disease, congestive heart failure, severe heart valve disease, acute myocarditis, acute and unstable musculoskeletal injuries, uncontrollable systemic hypertension, severe dementia and behavioral disorders)

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
FVC (Forced vital capacity ),%FVC | 12 weeks
  FVC was evaluated using a spirometer. The spirometer measurement results are compared FVC values with the expected values (predicted values) pre-calculated in healthy individuals of the same age, height and gender by the software found in the spirometer device and expressed as a percentage of these values.The results are delivered to the researcher by the authorised representative of the spirometer in pdf format within 15 days.
FEV1 (air volume after 1 second of forced expiration),%FEV1 | 12 weeks
  FEV1 was evaluated using a spirometer. The spirometer measurement results are compared FEV1 values with the expected values (predicted values) pre-calculated in healthy individuals of the same age, height and gender by the software found in the spirometer device and expressed as a percentage of these values. The results are delivered to the researcher by the authorised representative of the spirometer in pdf format within 15 days.
FEV1/FVC, %FEV1/FVC | 12 weeks
  FEV1/FVC was evaluated using a spirometer. The spirometer measurement results are compared FEV1/FVC with the expected values (predicted values) pre-calculated in healthy individuals of the same age, height and gender by the software found in the spirometer device and expressed as a percentage of these values.The results are delivered to the researcher by the authorised representative of the spirometer in pdf format within 15 days.

SECONDARY OUTCOMES:
Systolic blood pressure | 12 weeks
  Systolic blood pressure was evaluated using a manual sphygmomanometer. Measurement results before and after the intervention are recorded by the researcher.
Diastolic blood pressure | 12 weeks
  Diastolic blood pressure was evaluated using a manual sphygmomanometer. Measurement results before and after the intervention are recorded by the researcher.
Heart rate | 12 weeks
  Heart rate was evaluated using a pulse oximeter, Measurement results before and after the intervention are recorded by the researcher.
Oxygen saturation | 12 weeks
  Oxygen saturation was was evaluated using a pulse oximeter, Measurement results before and after the intervention are recorded by the researcher.
Pittsburgh Sleep Quality Index (PSQI) | 12 weeks
  The PSQI contains 18 self-rated questions and measures the quality of sleep over the last 4 weeks. The total score ranges from 0 to 21. An overall score higher than 5 indicates poor quality of sleep. The Cronbach α internal consistency coefficient of the scale is 0.80.
Subjective Vitality Scale (SVS) | 12 weeks
  The SVS is a 7-point Likert-type instrument with 7 self-rated items. The total score of the scale ranges from 7 to 49. A higher score indicates a higher level of subjective vitality. The Cronbach α internal consistency coefficient of the scale is 0.87.

CONTACTS AND LOCATIONS:
Overall Officials: Naile Bilgili, Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study method can be explained. Results will be shared after the study is published

REFERENCES:
- [Result] Jansang S, Mickleborough T, Suksom D. Effects of Pursed-Lip Breathing Exercise Using Windmill Toy on Lung Function and Respiratory Muscle Strength in the Elderly. J Med Assoc Thai. 2016 Sep;99(9):1046-51. PMID 29927211
- See also: World Health Organization. Top 10 causes of death. — http://www.who.int/news-room/fact-sheets/detail/the-top-10-causes-of-death#:~:text=The%20top%20global%20causes%20of,birth%20asphyxia%20and%20birth%20trauma%2C

DOCUMENTS (3):
  • Study Protocol (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04469972/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04469972/SAP_001.pdf
  • Informed Consent Form (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04469972/ICF_002.pdf